CLINICAL TRIAL: NCT00403052
Title: Phase 1 Study of the Combination of 1018 ISS, Irinotecan and Cetuximab in Patients With Metastatic Colorectal Cancer Previously Treated With a Fluoropyrimidine, Oxaliplatin or Irinotecan With or Without Bevacizumab
Brief Title: A Study of 1018 Immunostimulatory Sequence (ISS) Administered With Irinotecan and Cetuximab to Treat Patients With Previously Treated Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Administrative reasons
Sponsor: Dynavax Technologies Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DV2-ONC-01
Record Dates: First submitted 2006-11-21; First posted 2006-11-23 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Colorectal Neoplasms
Keywords: colorectal; cancer; carcinoma; metastatic; colon; rectal; neoplasm; cetuximab; irinotecan; 1018 ISS; combination therapy
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms; Carcinoma; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Low dose of 1018 ISS
  Interventions: Drug: 1018 ISS immunostimulatory oligonucleotide
- 2 (Experimental): Middle dose of 1018 ISS
  Interventions: Drug: 1018 ISS immunostimulatory oligonucleotide
- 3 (Experimental): High dose of 1018 ISS
  Interventions: Drug: 1018 ISS immunostimulatory oligonucleotide

INTERVENTIONS:
Drug: 1018 ISS immunostimulatory oligonucleotide — 6 weekly subcutaneous (under the skin) injections

SUMMARY:
The main objectives of this study are to establish a safe, tolerable and active dose of 1018 ISS administered in combination with irinotecan and cetuximab in patients with metastatic colorectal cancer. Other objectives also include determining tumor response, time to disease progression, and overall survival in treated patients.

DETAILED DESCRIPTION:
This is a Phase I, open-label study of escalating dose levels of 1018 ISS in combination with irinotecan and cetuximab in patients with previously treated metastatic colorectal cancer. Approximately 15 patients will be treated. The objectives of this study are to establish a safe, tolerable, and active dose of 1018 ISS, determine tumor response, time to disease progression, and overall survival in treated patients.

The safety and tolerability of 1018 ISS will be evaluated by periodic laboratory assessments, physical examinations, and compilation of adverse events.

Once study patients have been consented, screened, and assigned to one of the dose levels of 1018 ISS, patients will receive two 4 week cycles of 1018 ISS therapy plus irinotecan every other week and cetuximab weekly. Irinotecan and cetuximab will continue thereafter until disease progression, unacceptable toxicity, or until the patient refuses treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed, written, informed consent must be obtained from the patient or their legal representative before any study-specific procedures are performed
* Confirmed diagnosis of adenocarcinoma of the colon or rectum not amenable to curative surgery
* One or more prior systemic therapy regimens for metastatic cancer which must have included a fluoropyrimidine (5-fluorouracil (FU) by infusion or capecitabine), oxaliplatin or irinotecan with or without bevacizumab

Exclusion Criteria:

* Clinically significant obstructive symptoms, intestinal bleeding, or chronic or recent acute gastrointestinal disorder with diarrhea as a major symptom
* History of unstable or deteriorating cardiovascular or cerebrovascular disease within 3 months before the first dose of protocol therapy
* Clinical evidence of brain metastases or central nervous system disease
* Pregnant or lactating women
* Serious medical or psychiatric illness
* Malignancy other than colorectal carcinoma within the past 2 years, except curatively treated, superficial skin cancer or carcinoma in situ of the cervix
* Patients who have been on any experimental study or anti-tumor therapy, received radiotherapy, or had prior surgery (except venous access device placement) within 28 days before the first dose of protocol therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2006-11; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events | 16 weeks

SECONDARY OUTCOMES:
Time to tumor progression | 9 or more weeks
Overall survival time | 9 or more weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Martins, MD, DPhil, Study Director — Dynavax Technologies Corporation
Locations (3):
- United States (3):
  - Premiere Oncology, Santa Monica, California
  - Lombardi Comprehensive Cancer Center, Georgetown University, Washington D.C., District of Columbia
  - Center for Cancer and Blood Disorders, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: Undecided
3/2017 No change in status of this study

REFERENCES:
- See also: Dynavax Webpage — http://www.dynavax.com